CLINICAL TRIAL: NCT04613973
Title: Evaluation of the Program to Help Return Home Patients Hospitalized for Heart Failure, in a Cohort of Patients From the Hôpital Paris Saint-Joseph
Brief Title: Evaluation of the Program to Help Return Home Patients Hospitalized for Heart Failure, From Paris Saint-Joseph Hospital
Acronym: PRADO_IC2
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PRADO_IC2
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients included in the PRADO program: Patients hospitalized for global heart failure or left ventricular insufficiency in the Cardiology department of the GHPSJ between January 2016 and September 2018, included in the support program for Return To Home for Heart Failure (PRADO)
- Patients not included in the PRADO program: Patients hospitalized for global heart failure or left ventricular insufficiency in the Cardiology department of the GHPSJ between January 2016 and September 2018, not included in the Return A DOmicile support program for Heart Failure (PRADO)

SUMMARY:
The prevalence of heart failure is very high worldwide is between 1 and 2% in developed countries.

The French Federation of Cardiology estimates that a million people are affected in France. Each year in France, there are nearly 70,000 deaths linked to heart failure, and more than 150,000 hospitalizations with an average cumulative duration per year of 12.7 days, figures which show the extent of the phenomenon. Heart failure is therefore a common pathology, which constitutes an important public health issue. It requires rigorous monitoring and early adaptation of treatments to avoid repeated hospitalizations. Studies show that following hospitalization for heart failure, all-cause re-hospitalization rates rise to 18% within 30 days. In 2019, the rate of re-hospitalization at 1 year is 30%, half of which in the following 3 months. The prognosis is grim with 20 to 30% of deaths within the year.

The European Society of Cardiology recommends that the patient be integrated into a care path coordinated by the general practitioner; and a consultation with his general practitioner in the week after hospitalization and his cardiologist within two weeks. The CPAM (Caisse Primaire d'Assurance Maladie) has set up since 2013 the PRADO-IC program (Program for Return to Home Hospital for Heart Failure). This program must be in place before discharge from hospital. A health insurance advisor comes to meet the patient, declared eligible for PRADO by the hospital medical team, to present the offer and collect his approval before discharge. He then contacts the attending physician and organizes his return home. A follow-up book is given to the patient to allow better transmission of information between town and hospital.

A specially trained nurse visits the patient's home every week. The duration of PRADO support varies according to the NYHA stage of severity. It provides therapeutic education with reinforcement of hygieno-dietetic rules, warning signs, checks compliance with treatments and the necessary biological monitoring and must alert the attending physician in the event of aggravation.

The objectives of this program are: to preserve the quality of life and the autonomy of patients, to support the reduction of the length of stay in hospital, to strengthen the quality of care in town around the attending physician, improve the efficiency of recourse to hospitalization by reserving the heaviest structures for the patients who need them most.

DETAILED DESCRIPTION:
The prevalence of heart failure is very high worldwide: according to the European Society of Cardiology, it is between 1 and 2% in developed countries.

The French Federation of Cardiology estimates that a million people are affected in France. This prevalence increases sharply with age, reaching 15% of people aged 85 and over.

Each year in France, there are nearly 70,000 deaths linked to heart failure, and more than 150,000 hospitalizations with an average cumulative duration per year of 12.7 days, figures which show the extent of the phenomenon. In addition, the aging of the population and the explosion of cardiovascular risk factors suggest that the impact of heart failure will be greater in the future.

Heart failure is therefore a common pathology, which constitutes an important public health issue. It requires rigorous monitoring and early adaptation of treatments to avoid repeated hospitalizations. Studies show that following hospitalization for heart failure, all-cause re-hospitalization rates rise to 18% within 30 days. According to a report from the Caisse Primaire d'Assurance Maladie (CPAM) in 2019, the rate of re-hospitalization at 1 year is 30%, half of which in the following 3 months. The prognosis is grim with 20 to 30% of deaths within the year.

The European Society of Cardiology recommends that the patient be integrated into a care path coordinated by the general practitioner; and a consultation with his general practitioner in the week after hospitalization and his cardiologist within two weeks. But general practitioners deplore a lack of coordination between city and hospital with difficulties in taking care of their patient following hospitalization. According to the CPAM report, only 30% of re-hospitalized patients had contact with a cardiologist before their readmission, and 15% of patients had no contact with the health care system within 2 months of followed their hospitalization.

It is in this need to improve monitoring that the CPAM has set up since 2013 the PRADO-IC program (Support Program for Return to Home Hospital for Heart Failure). This program must be in place before discharge from hospital. A health insurance advisor comes to meet the patient, declared eligible for PRADO by the hospital medical team, to present the offer and collect his approval before discharge. He then contacts the attending physician and organizes his return home. A follow-up book is given to the patient to allow better transmission of information between town and hospital.

A specially trained nurse (internet training) visits the patient's home every week. The duration of PRADO support varies according to the NYHA stage of severity: a patient in NYHA stage I or II benefits from home support for a period of 2 months, and 6 months for NYHA stages III and IV. It should make it possible to monitor the constants: blood pressure, pulse, and weight. It provides therapeutic education with reinforcement of hygieno-dietetic rules (low sodium diet), warning signs (orthopnea, cough, dyspnea), checks compliance with treatments and the necessary biological monitoring and must alert the attending physician in the event of aggravation.

The objectives of this program are: to preserve the quality of life and the autonomy of patients, to support the reduction of the length of stay in hospital, to strengthen the quality of care in town around the attending physician, improve the efficiency of recourse to hospitalization by reserving the heaviest structures for the patients who need them most.

The main objective of this study is therefore to assess the impact of the PRADO program on re-hospitalization at 1 year, at Paris Saint-Joseph hospital for heart failure.

ELIGIBILITY:
Inclusion Criteria:

Patients included in PRADO

* Patient whose age is ≥ 18 years
* Patient hospitalized for global heart failure or left ventricular failure in the Cardiology department of the GHPSJ between January 2016 and September 2018
* Patients included in the PRADO program Patients not included in PRADO
* Patient whose age is ≥ 18 years
* Patient hospitalized for global heart failure or left ventricular failure in the Cardiology department of the GHPSJ between January 2016 and September 2018
* Patients not included in the PRADO program

Exclusion Criteria:

* Patient under guardianship or guardianship
* Patient living in EHPAD
* Patient transferred to another establishment on discharge from hospital (surgery, follow-up care, EPHAD, etc.)
* Patient who died during hospitalization
* Patient objecting to the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for global heart failure or left ventricular failure in the Cardiology department of the GHPSJ between January 2016 and September 2018.
Sampling Method: Non-Probability Sample
Enrollment: 633 (Actual)
Dates: Start 2020-11-28 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Impact of the PRADO program on re-hospitalization at 1 year | Year 1
  This outcome corresponds to 1-year re-hospitalization rate for heart failure after an episode of cardiac decompensation in patients included in the PRADO program vs. patients not included in PRADO.

SECONDARY OUTCOMES:
Mortality at 1 year | Year 1
  This outcome corresponds to the mortality at 1 year.
First re-hospitalization | Year 1
  This outcome corresponds to the delay until the first re-hospitalization during the year.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ABASSADE, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Tuppin P, Cuerq A, de Peretti C, Fagot-Campagna A, Danchin N, Juilliere Y, Alla F, Allemand H, Bauters C, Drici MD, Hagege A, Jondeau G, Jourdain P, Leizorovicz A, Paccaud F. First hospitalization for heart failure in France in 2009: patient characteristics and 30-day follow-up. Arch Cardiovasc Dis. 2013 Nov;106(11):570-85. doi: 10.1016/j.acvd.2013.08.002. Epub 2013 Oct 18. PMID 24140417
- [Result] Assyag P, Renaud T, Cohen-Solal A, Viaud M, Krys H, Bundalo A, Michel PL, Boukobza R, Bourgueil Y, Cohen A. RESICARD: East Paris network for the management of heart failure: absence of effect on mortality and rehospitalization in patients with severe heart failure admitted following severe decompensation. Arch Cardiovasc Dis. 2009 Jan;102(1):29-41. doi: 10.1016/j.acvd.2008.10.013. Epub 2009 Feb 10. PMID 19233107
- [Result] Desai AS. The three-phase terrain of heart failure readmissions. Circ Heart Fail. 2012 Jul 1;5(4):398-400. doi: 10.1161/CIRCHEARTFAILURE.112.968735. No abstract available. PMID 22811548
- [Result] Abassade P, Cohen L, Fels A, Chatellier G, Sacco E, Beaussier H, Fleury L, Komajda M, Cador R. [Impact of Home Return Assistance Service in Heart Failure (PRADO-IC) on the one year re-hospitalisation and mortality in a heart failure hospitalized population of patients]. Ann Cardiol Angeiol (Paris). 2022 Nov;71(5):267-275. doi: 10.1016/j.ancard.2022.07.004. Epub 2022 Aug 6. French. PMID 35940973